CLINICAL TRIAL: NCT04984200
Title: Assessment of EyeArt Performance With Retinal Cameras
Status: Completed | Type: Observational
Sponsor: Eyenuk, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EN-01b
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Mydriatics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- AB
  Interventions: Procedure: Retinal imaging; Drug: Mydriatic Agent

INTERVENTIONS:
Procedure: Retinal imaging — Subjects will undergo retinal imaging before and/or after administration of mydriatic agent
Drug: Mydriatic Agent — Subjects will be administered mydriatic medication to dilate their pupils.

SUMMARY:
The study evaluates the performance of the EyeArt system for detecting diabetic retinopathy from images captured using retinal cameras and operators.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of diabetes mellitus;
* Understanding of study and provision of written informed consent; and
* 22 years of age or older.

Exclusion Criteria:

* Persistent visual impairment in one or both eyes;
* History of retinal vascular (vein or artery) occlusion;
* History of ocular injections, laser treatment of the retina, or intraocular surgery other than cataract surgery without complications;
* Subject is contraindicated for fundus photography (for example, has light sensitivity);
* Subject has contraindications for mydriatic medications or is unwilling or unable to dilate;
* Subject is currently enrolled in an interventional study of an investigational device or drug; or
* Subject has a condition or is in a situation which in the opinion of the Investigator, might confound study results, may interfere significantly with the subject's participation in the study, or may result in ungradable dilated fundus photographs.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be enrolled at primary care and/or eye care centers
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Overall agreement between the results from multiple EyeArt operations | 1 visit (1 day)
  Overall agreement is defined as the fraction of cases where the multiple EyeArt operation results agree with each other.

CONTACTS AND LOCATIONS:
Locations (1):
- Rocky Mountain Diabetes Center, Idaho Falls, Idaho, United States